CLINICAL TRIAL: NCT02727127
Title: Brain Ion Homeostasis, Lithium and Bipolar Disorder
Status: Terminated | Type: Observational
Why Stopped: Lost funding due to low enrollment
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 12-03629
Record Dates: First submitted 2016-03-29; First posted 2016-04-04 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Healthy; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Volunteers: MRI on 3 Tesla (3T) or 7 Tesla (7T) scanner, without contrast
- Bipolar Patients: MRI on 3 Tesla (3T) or 7 Tesla (7T) scanner, without contrast

SUMMARY:
In this project, investigators intend to carry out the first simultaneous, in vivo, imaging study of lithium content and sodium ion homeostasis in the brain of Bipolar Disorder (BPD) patients under Lithium therapy.

DETAILED DESCRIPTION:
The purpose of this study is to validate a new method for the measurement of the amount of lithium (also known as lithium concentration) in the brain of subjects undergoing lithium treatment for bipolar disorder. The method involves the use of Magnetic Resonance Imaging (MRI) and Spectroscopy (MRS) techniques. These are non-invasive techniques, with no known harmful effects, that allow investigators to measure the amount of lithium in an individual's brain. There will be no contrast dye used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatrically stable patients (diagnosed according to the Diagnostic and Statistical Manual, DSM-IV, criteria)
* On steady state serum lithium levels (0.8-1.2mEq/L)

Exclusion Criteria:

* Subjects who have a history of head trauma
* Subjects who have a contraindication for an MRI exam, including a claustrophobia, surgical or vascular implants, pregnancy, pacemakers, neurostimulators, history of metal in the eyes, and orthodontia or extensive bridgework (with have a particular impact on gradient echo imaging).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of New York City and surrounding areas
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-09; Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Study the relationship between BLC and brain sodium ion homeostasis, as measured by concurrent Single / Triple quantum sodium MRI in BPD patients | 1 Hour

SECONDARY OUTCOMES:
To investigate the measurement of sodium ion homeostasis in the brain of BPD patients, at clinical magnetic field strengths (3 Tesla), as a non-invasive surrogate marker of BLC during Lithium Carbonate therapy | 1 Hour

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Boada, PhD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No